CLINICAL TRIAL: NCT00232843
Title: A Clinical Investigation of the SMART™ Nitinol Self-Expandable Stent Versus Balloon Angioplasty Only for the Treatment of SUPERficial Femoral Artery Occlusions
Brief Title: The Study to Treat Superficial Femoral Artery Occlusions.
Acronym: SUPER UK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EE04-01UK
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Arterial Occlusive Diseases
Keywords: Peripheral Artery Occlusive Disease
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Arterial Occlusive Disease 1 | interventions — Stents; Angioplasty; Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cordis SMART™ nitinol self-expanding stent.
  Interventions: Device: stent
- 2 (Active Comparator): balloon angioplasty
  Interventions: Device: angioplasty

INTERVENTIONS:
Device: stent — Cordis SMART™ nitinol self-expanding stent.
  Other Names: Cordis SMART™ nitinol self-expanding stent
  Arms: 1
Device: angioplasty — balloon angioplasty
  Other Names: balloon angioplasty
  Arms: 2

SUMMARY:
The main objective of this study is to assess the performance of the Cordis SMART™ nitinol self-expandable stent for the treatment of superficial femoral artery (SFA) occlusions in comparison with balloon angioplasty only as determined by binary restenosis at one year.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, two-arm study evaluating the performance of the Cordis SMART™ nitinol self-expanding stent as compared to angioplasty only.

It is anticipated that a total of 150 patients will be entered into the study. Patients will be randomized on a 1:1 basis of stent versus angioplasty only.

150 patients with de novo or restenotic native SFA occlusions (5-22 cm) with reference vessel of >= 4.0 to <= 6.0 mm in diameter will be randomized to the SMART™ nitinol self-expanding stent or to angioplasty only.

All patients will be followed for 12 months post-procedure, by telephone contact at 3 and 6 months, and a 12 month clinical and duplex ultrasound assessment. This study will be conducted at up to 12 investigational sites.

ELIGIBILITY:
Inclusion Criteria:

* One superficial femoral artery de novo or restenotic lesion (> 70% stenosis or occlusions), with a lesion length > 5 to < 22 cm.
* Patent popliteal artery on the index side, i.e., single vessel runoff or better with at least one of three vessels patent to the lower 1/3 of the calf prior to the day of the procedure. Additional intervention to further improve blood flow to the lower limb is acceptable during the index procedure, but after successful treatment of the study lesions

Exclusion Criteria:

* Revascularisation involving the same limb within 7 days prior to the index procedure or a planned revascularisation within 7 days after the index procedure Patient having total occlusions of the iliac artery on the same side must be excluded. However, intervention to restore adequate blood flow is allowed during the same procedure and prior to the treatment of the study lesion.
* Patients enrolled in this or other clinical trial or anticipated to be included into a trial, without written approval of the Cordis medical monitor and the principal investigator of this study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Binary restenosis as demonstrated by Duplex Ultrasound. | 1 year

SECONDARY OUTCOMES:
Device success. | at time of deployment
Procedural success: defined as successful recanalization, without the occurrence of a SAE event. | up to the moment the catheter sheath introducer has been removed
Ankle Brachial Index | at discharge and 12 months
Restenosis measured by Duplex Ultrasound | at discharge and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nick Chalmers, MD, Principal Investigator — Manchester Royal Infirmary; Mark Cowling, MD, Principal Investigator — University Hospital of North Staffordshire
Locations (2):
- United Kingdom (2):
  - Manchester Royal Infirmary, Manchester
  - University Hospital of North Staffordshire, Newcastle-under-Lyme